CLINICAL TRIAL: NCT03249649
Title: Enhancing Culturally-Informed Health Care Services for Women Affected by Female Genital Cutting in Arizona
Brief Title: Female Genital Cutting in the Arizona Somali Refugee Community
Acronym: FGC
Status: Completed | Type: Observational
Sponsor: Arizona State University (Other)
Collaborators: Catholic Charities (Other); Phoenix International Refugee Committee (Unknown); Refugee Focus Phoenix (Unknown); Refugee Focus Tucson (Unknown); Somali Bantu Community of Greater Phoenix (Unknown); Horizons Refugee Families (Unknown)
Responsible Party: Principal Investigator, Crista Johnson-Agbakwu, Principal Investigator, Arizona State University
Other Study IDs: 5252
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Female Genital Mutilation Type I Status; Female Genital Mutilation Type II Status; Female Genital Mutilation Type III Status
Keywords: defibulation; healthcare needs assessment; CBPR

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phoenix Cohort: Somali Refugee women ages 15 and older
  Interventions: Behavioral: Comprehensive Healthcare Needs Assessment
- Tucson Cohort: Somali Refugee women ages 15 and older
  Interventions: Behavioral: Comprehensive Healthcare Needs Assessment

INTERVENTIONS:
Behavioral: Comprehensive Healthcare Needs Assessment — Questionnaire focused on existing healthcare communication, treatment and services plus community needs in those three areas.

SUMMARY:
The focus of this project is to elucidate the gaps in care and enhance the provision of FGC-related health care and social services for women in Arizona who have experienced FGC; engaging the Somali and Somali Bantu communities. As of 2012, Arizona ranked 7th in the US for Somali refugee resettlement. The Refugee Women's Health Clinic (RWHC) is a nationally recognized best practice model for refugee women's health, providing specialized care for women with FGC. The project will accomplish four outcomes throughout its three-year duration: 1: Identify specific FGC-related health care needs and available health and social services for women in Arizona who have experienced FGC to improve services to FGC-affected communities; 2: Identify gaps, barriers, and/or assets in FGC-related health care and social services for women in Arizona who have experienced FGC to provide improved services to FGC-affected communities; 3: Create and implement FGC education efforts so that providers improve culturally competent care for women who have experienced FGC in health care and social service settings; and, 4: Create and implement community outreach and educational programs among communities affected by FGC to increase awareness of FGC-related health issues, prevention and services available. To inform these initiatives, an established infrastructure exists through the Refugee Women's Health Community Advisory Coalition (RWHCAC), a team of more than 60 stakeholders from various local ethnic organizations, refugee resettlement and voluntary agencies, mental health and social services agencies, and academic partners and including local voluntary resettlement agencies (VOLAGs) and Ethnic Community-Based Organizations (ECBOs). RWHCAC will be (a) involved in the planning/design of the project, (b) encouraged to assume responsibility to identify additional Community Mobilizers, (c) engaged in aligning educational material content to cultural standards, and (d) engaged in evaluating the project processes and outcomes.

Project strategies include: (1) identifying specific FGC-related health care needs and available health and social services for FGC-affected women including identification of gaps, barriers, and/or assets in FGC-related care (year 1); (2) utilizing results from the Community Health Needs Assessment (CHNA) to refine existing educational materials and implement educational outreach efforts across the state to improve culturally competent care among providers (years 2 and 3); (3) promoting outreach and education among FGC-affected communities through development of culturally appropriate materials and community education sessions (years two and three); and, (4) partnering with Arizona Department of Health Services, the University of Arizona, and African Women's Health Center, Brigham and Women's Hospital during year 2 to deliver inter-professional training workshops for health and social service providers on FGC, and with Johns Hopkins University for FGC teleECHO™ video conferencing clinics to promote sustainability via links to online resources, educational materials, and webinars (years 2 and 3). Emergent products include online learning components, community education sessions, FGC teleECHO™ sessions, and capacity building trainings for all partners.

DETAILED DESCRIPTION:
Prevalence of Female Genital Cutting (FGC) in Arizona is uncertain; no available state or national surveys with either prevalence or risk estimates exist, necessitating estimates indirectly derived. Acknowledging a diversity of African-born communities where FGC is prevalent within Arizona, for this proposal our team chose to focus specifically on the Somali and Somali Bantu communities in Phoenix and Tucson for three reasons: 1) size of the community and FGC-related health care concerns, 2) Type III FGC (most severe form) is most common among Somali women, and 3) a long-standing record of robust community partnerships that exist among our partnering agencies and the Somali community. This Project Community will establish comprehensive strategies to ensure diverse input from partners in developing collaborative operating principles. The community partners will be: 1) involved in the planning and design of the project; 2) given the responsibility to identify Community Mobilizers; and, 3) evaluate and align the educational content of outreach materials to match cultural standards.

RWHC Clinical Care, Prior Research, and History of CBPR Engagement/Partnership RWHC: Since 2008, RWHC at Maricopa Integrated Health System (MIHS) has addressed disparities in knowledge and expertise in care of women with FGC, establishing a patient-centered medical home for refugee women. The first of its kind in Arizona, it is nationally recognized as a best practice model for refugee women's health care, addressing reproductive health disparities among newly-resettled refugee women. The multilingual, bicultural staff, refugee women who serve as Cultural Health Navigators (CHNs), facilitate an integrated team approach to comprehensive health care delivery and health care system navigation. RWHC has robust partnerships with local communities affected by FGC, engaging in Community-Based Participatory Research (CBPR) to enhance community collaboration in culturally relevant intervention/program design. Despite these efforts, there remains a critical need for increased provider cultural competency in caring for FGC-affected populations and in de-monopolizing care so that providers become skilled in caring for FGC-affected women.

Prior Research: Training among Healthcare Providers: In 2014, RWHC surveyed 508 US healthcare providers to assess awareness of FGC, prior training exposure, and current approaches to care for women affected by FGC. Results showed widespread knowledge gaps among providers, with 81% expressing a desire for further education/training on FGC. Results also showed that exposure to FGC training and direct clinical care encounters with FGC-affected populations predicted increased competency in the care of these women.

Prior Research: Gaps between Providers and Somali Women: Our team conducted a mixed-methods study in Maricopa County, Arizona (July 2011-May 2012) exploring knowledge, perceptions and experiences in the context of FGC among Somali women (n=73) and obstetrics/gynecology healthcare providers (n=74). Findings suggested a substantial lack of agreement between Somali women and health care providers on prenatal care, labor, and delivery in the context of FGC. Although providers often failed to recognize FGC-related health concerns and management around childbirth and agreed they lacked formal training on FGC- related care, they linked all types of FGC to adverse birth outcomes. Stigmatization, alienation, distrust, lack of cultural knowledge and clinical skills, and fear of surgical interventions led Somali women to delay prenatal care and arrangements for labor and delivery while they categorically rejected the imposed construct of "FGC-victimization." History of Community Engagement/Partnership: An established infrastructure of community partnership, engagement, and shared community leadership exists through the Refugee Women's Health Community Advisory Coalition (RWHCAC). The RWHCAC is an interdisciplinary team of more than 60 stakeholders from various community organizations representing local ethnic organizations, refugee resettlement and volunteer agencies, mental health and social services agencies, and academic partners. Through RWHCAC, we have partnered with the Somali community on numerous collaborative initiatives to build community capacity on Somali reproductive health issues of importance Goal and Anticipated Outcome To address health disparities for Somali women, the goal of this initiative will be to elucidate gaps in care and enhance the provision of FGC-related health care and social services for women in Arizona who have experienced FGC. Outcome 1: Identify specific FGC-related health care needs and available health and social services for FGC-affected women in Arizona. Outcome 2: Identify gaps, barriers, and/or assets in FGC-related health care and social services for women in Arizona. The Somali community has expressed their desire for greater engagement of all community stakeholders in providing community-wide education enhancing community awareness on available health services/resources, interpreting FGC-related legislation, and educating health care providers. Outcome 3: Create and implement FGC education efforts to improve culturally competent care in healthcare and social service settings for FGC-affected women. Outcome 4: Implement comprehensive community outreach and education about FGC- related health issues, prevention, and services available.

Year 1 Strategy: Outcomes 1 and 2 will be addressed by identifying specific FGC-related health care needs and available health and social services for FGC-affected women including an identification of the gaps, barriers, and/or assets in FGC-related care. Instrument: The CNHA will assess baseline and interval changes in: knowledge, attitudes, and behavioriii on FGC-health related issues, as well as gaps, barriers and/or assets in the receipt of health services (see Work Plan Appendix). This same survey will re-administered in-person or via telephone by Community Mobilizers in Year 3 to assess changes in knowledge, attitudes and behavior.

Recruitment: A Respondent-Driven Sampling (RDS) strategy will be used to recruit community participants in this project. RDS is an effective method for recruiting "hidden" populations, such as refugee populations and when participant behaviors are stigmatized. The RDS is an advanced adaptation of the traditional snowball sampling method; a small number of selected initial recruiters (socially connected community mobilizers and organizations) generate a list of potential recruits from their social networks, connections and community memberships. They are given distinctive identifying coded coupons and incentives to create the first wave of recruits. The first wave of recruits will also be incentivized to recruit a second wave, and so on; the wave after wave recruitment cycle will continue until equilibrium is attained and sample size is achieved. We performed a precision analysis to estimate a sample size based on the prevalence rate of FGC in the population, the margin of error desired, the confidence interval, the total population size, the expected attrition, and the design effect from using RDS. We expect 40 percent attrition, with a population size of about 3,300 women, and a RDS design effect of 2, thus a need to retain 2,040 women in the sample. Data Management: Each questionnaire will be given a unique identifier code to match coded coupons of the community mobilizer to identify the specific wave it originated from. Data entry will occur in the field, completed by surveyors, eliminating the need for further entry processes so that preliminary analyses will proceed concurrently. CHNA results will inform the educational training among health and social service providers as well as community educational outreach for providers and community members.

Barriers and Assets: Potential barriers include low literacy, trust, confidentiality, ethnic/clan affiliation, and/or discussion of FGC as a sensitive/taboo subject matter. To address these concerns, the survey will be verbally administered in Somali and/or Maay Maay by female Community Mobilizers sharing the same ethnic/cultural/linguistic background as the participant. Community Mobilizers, trained on human subjects protections regarding consent and confidentiality, will conduct interviews in settings deemed appropriate and safe by the participant, and in respect for Muslim prayer times.

Year 2 - 3 Strategy: Utilizing CHNA results we will refine and implement educational outreachefforts across the state to improve provider culturally competent care of FGC-affected women and to promote community education about the prevention of FGC. Health care and Provider Education: A detailed description of partnerships for provider education and training in Year 2 are included in the Work Plan Appendix. Sustainability: Throughout Years 2 and 3, participants in the workshops will be invited to join FGC ECHO, through monthly FGC teleECHO™ video conferencing clinics. This educational outreach will build culturally competent care expertise across a wider net of health and social service providers to improve health outcomes. Providers will be offered links to online educational resources and webinars, and ADHS BWCH/RHP will offer continuous support. Bridging Refugee Youth and Children's Services (BRYCS), a current Office of Refugee Resettlement (ORR)-funded technical assistance (TA) provider, will enhance efforts through its website, national Clearinghouse and newsletters across a diverse platform of providers. Data Management: Pre-post surveys will be conducted at baseline, Year 2, and 15 months after the workshop completion in Year 3. Analyses will assess changes in provider knowledge, attitudes towards FGC, and clinical care and management. Barriers and Assets: To address the potential for low provider attendance at the educational workshops, we will offer Continuing Medical Education/Continuing Education Unit (CME/CEU) credits to promote provider professional development, and specifically, to target providers and health care institutions serving FGC-affected communities. Assets that will ensure strong provider attendance and sustainable access to professional development are ADHS BWCH/RHP's resources to host live webinars for those who are unable to attend the workshops in-person.

BRYCS will facilitate statewide and national dissemination of provider educational materials through its online network of 7,000+ members and strong social media following. Benefits to other communities: Arizona will be one of 10 states participating in the provider workshops led by Dr. Nawal Nour. Data gathered from pre-post surveys will inform national efforts to address gaps in provider and community knowledge. Furthermore, the FGC ECHO initiative promises far-reaching implications for improving provider competency and skill in regions where there are no FGC specialists. Specific products/outcomes proposed for development or modification beyond the OWH final report: Providers will receive a workshop program workbook on caring for FGC-affected populations, links to online resources, webinars and ongoing access to FGC, ECHO and BRYCS networks of inter-professional providers. Community Outreach and Education: Prior collaborations have demonstrated the critical role of men in women's healthcare decision-making. Moreover, cultural etiquette requires male forums to be held separately from female forums. Community forums will be convened and led by trained community leaders and will break into small groups organized by generational status comprising youth, elders, and the middle-aged to facilitate further discussions to illuminate specific community needs and educational priorities for providers (see Work Plan for details). During the FGC Listening Sessions held in 2014, the Somali community voiced a need to hear from religious leaders who could interpret the significance of FGC through the lens of their faith. In response to this request, leaders from the Islamic community will be invited to address the forums on FGC from a religious perspective. In particular, the forums will invite younger Somali women to address health care needs of women engaging in FGC and attitudes about prevention. Also, during the women's forums, participants will view the ORR Somali health educational video on FGC and receive a bilingual educational brochure on FGC to facilitate the empowerment of women to discuss their FGC-related care and management with their providers.

In Year 3, a follow-up CHNA will be re-administered. Community Mobilizers will conduct the surveys either in-person or via telephone. Role of Sub-recipients: One sub-recipient will provide support for additional time for the Project Lead and a Project Manager (see subcontract scope of work for details). Data Management: The Work Plan Appendix includes a detailed description of the tasks, performance measures and expected products from the community forums. Sustainability: This project will build capacity for Community Mobilizers, ECBOs and Community Representatives to be closely engaged with ongoing efforts of the VOLAGs, healthcare institutions, and RWHC/SIRC to promote refugee community health.

Strength and Expertise of the Applicant and Partnerships of Project Community: Project Lead, Dr. Crista Johnson-Agbakwu, MD, MSc, Founding Director of RWHC, brings nearly two decades of experience with FGC-affected communities. Her academic research home, the Southwest Interdisciplinary Research Center (SIRC) at Arizona State University, is anNIH/NIMHD Exploratory Center of Excellence in CBPR-driven health disparities research to address social and cultural processes as factors in the reduction and elimination of health disparities (P20MD002316). SIRC provides research infrastructure support including methods expertise, data management, statistical, grant development, and evaluation. As part of SIRC, the Project Lead guided a refugee health literacy demonstration project in partnership with RWHCAC. Thus, the RWHC/SIRC partnership is well-positioned to co-lead this project. The Project Community, comprised of members of the RWHCAC including local voluntary resettlement agencies (VOLAGs), Ethnic Community-Based Organizations (ECBOs), individual Somali/Somali Bantu Community Representatives, and local health care institutions in Phoenix and Tucson, has been engaged in planning this proposal and will be immersed in all phases of implementation, reporting, statewide dissemination and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* live and receive healthcare treatment and social services in Arizona
* meet the age criteria

Exclusion Criteria:

* males
* non-Somali Refugee women

Min Age: 15 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Somali and Somali Bantu Refugee females ages 15 and older
Study Population: Somali and Somali Bantu Refugee females ages 15 and older who have been resettled to Arizona and who have received healthcare, health services, and/or social services from Arizona providers.
Sampling Method: Non-Probability Sample
Enrollment: 1736 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Comprehensive Healthcare Needs Assessment (CHNA) | 7/1/2016-12/31/2017
  Measure of patient-provider communication, patient healthcare services, and provider treatment of Somali Refugee women.
Gaps, Barriers, and Assets in FGC Related Healthcare | 1/1/2018-6/30/2018
  Report on gaps, barriers, and/or assets in FGC-related health care and social services for women in Arizona.
Provider Education and Training | 7/1/2018-6/30/19
  Report on FGC education efforts to improve culturally competent care in healthcare and social service settings for FGC-affected women.
Community Education and Training | 7/1/2018-6/30/19
  Report on comprehensive community outreach and education about FGC- related health issues, prevention, and services available.

CONTACTS AND LOCATIONS:
Overall Officials: Crista Johnson-Agbakwu, MD, Principal Investigator — Arizona State University
Locations (1):
- Southwest Interdisciplinary Research Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available for use by qualified individuals within the scientific community after publication. The quantitative data will be made available in SPSS (.sav format), after removing from the file any information personally identifying human subjects. A codebook, produced in SPSS, and a brief summary of the original study, including information on sampling and design, will accompany the dataset. Qualitative data that contain no identifiers will be made available in text files (.txt format). Requests for the data will be made in writing directly to the principal investigator. Requestors must indicate the research question to be addressed. Users will not be permitted to share the requested data with other users unless they have the express permission of the principal investigator. Users' acknowledgement of these requirements will be recorded in a signed Use Agreement, to be kept on file at the principal investigator's offices.
Supporting Information: Analytic Code
Time Frame: Data will become available following publication of all manuscripts reporting outcomes of primary and secondary aims. It is anticipated that these data will be available beginning year 7 and for 7 years following.
Access Criteria: Access criteria are identified in the plan to share IPD.

REFERENCES:
- [Derived] Johnson-Agbakwu CE, Michlig GJ, Koukoui S, Akinsulure-Smith AM, Jacobson DS. Health outcomes and female genital mutilation/cutting: how much is due to the cutting itself? Int J Impot Res. 2023 May;35(3):218-227. doi: 10.1038/s41443-022-00661-6. Epub 2023 Jan 4. PMID 36599966
- [Derived] Johnson-Agbakwu CE, Fox KA, Banke-Thomas A, Michlig GJ. Influence of Female Genital Mutilation/Cutting on Health Morbidity, Health Service Utilization and Satisfaction with Care among Somali Women and Teenage Girls in the United States. J Racial Ethn Health Disparities. 2023 Apr;10(2):788-796. doi: 10.1007/s40615-022-01266-x. Epub 2022 Mar 8. PMID 35258838
- [Derived] Marea CX, Warren N, Glass N, Johnson-Agbakwu C, Perrin N. Assessing the reliability and validity of attitudes and confidence scales for the care of women and girls affected by female genital mutilation/cutting. BMC Public Health. 2021 Jul 17;21(1):1415. doi: 10.1186/s12889-021-11455-8. PMID 34273951
- [Derived] Marea CX, Warren N, Glass N, Johnson-Agbakwu C, Perrin N. Factors Associated with Health Care Provider Attitudes, and Confidence for the Care of Women and Girls Affected by Female Genital Mutilation/Cutting. Health Equity. 2021 May 19;5(1):329-337. doi: 10.1089/heq.2020.0130. eCollection 2021. PMID 34036217